CLINICAL TRIAL: NCT03545074
Title: Efficacy of Spanish or English Language Versions of Mindfulness Meditation on Depression: A Randomized Controlled Trial in Spanish or English Speaking Cohorts
Brief Title: Efficacy of Spanish or English Language Versions of Mindfulness Meditation on Depression
Acronym: REMAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Eric Lopez, PhD, Postdoctoral Fellow, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMAPS
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Depression
Keywords: mindfulness; depression; Spanish
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Pretest and immediate postest design with an active control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness Spanish (Experimental): The MAPs program was developed at UCLA (Winston & Smalley, 2010 and Lopez-Maya, 2016) and provides experiential training in mindfulness-based practices, including mindfulness meditation. UCLA-certified instructors delivered the interventions. Active program components include sitting and walking meditations, body scan and loving-kindness meditation. Participants were provided with audio CDs or digital downloads to complete their daily meditation assignments. Sessions were held once per week for 2 hours per session over a period of six consecutive weeks. Home practice assignments consist of daily mindfulness exercises starting with 5 minutes daily, progressing to 20 minutes daily by the end of the program.
  Interventions: Behavioral: Mindful Awareness Practices- Spanish
- Mindfulness English (Experimental): The MAPs program was developed at UCLA (Winston & Smalley, 2010) and provides experiential training in mindfulness-based practices, including mindfulness meditation. UCLA-certified instructors delivered the interventions. Active program components include sitting and walking meditations, body scan and loving-kindness meditation. Participants were provided with audio CDs or digital downloads to complete their daily meditation assignments. Sessions were held once per week for 2 hours per session over a period of six consecutive weeks. Home practice assignments consist of daily mindfulness exercises starting with 5 minutes daily, progressing to 20 minutes daily by the end of the program.
  Interventions: Behavioral: Mindful Awareness Practices- English
- Health Education Spanish (Active Comparator): The health education condition is a weekly 2-hour, 6 session course aimed at knowledge acquisition in subjects related to health care in general. Similar interventions have been described elsewhere (Black, et al., 2014; Irwin, et al., 2014). A trained health educator provided videos and didactic presentations on topics such as: stress, sleep hygiene, diet & nutrition, sexuality, mental health and substance abuse. The health education condition resembled the MAPs intervention in terms of duration, group format and support, attention and participant expectancy regarding health benefits.
  Interventions: Behavioral: Health Education - Spanish
- Health Education English (Active Comparator): The health education condition is a weekly 2-hour, 6 session course aimed at knowledge acquisition in subjects related to health care in general. Similar interventions have been described elsewhere (Black, et al., 2014; Irwin, et al., 2014). A trained health educator provided videos and didactic presentations on topics such as: stress, sleep hygiene, diet & nutrition, sexuality, mental health and substance abuse. The health education condition resembled the MAPs intervention in terms of duration, group format and support, attention and participant expectancy regarding health benefits.
  Interventions: Behavioral: Health Education - English

INTERVENTIONS:
Behavioral: Mindful Awareness Practices- English — The 6-week intervention aimed at teaching mindfulness-based strategies to participants (in English)
  Arms: Mindfulness English
Behavioral: Mindful Awareness Practices- Spanish — The 6-week intervention aimed at teaching mindfulness-based strategies to participants (in Spanish)
  Arms: Mindfulness Spanish
Behavioral: Health Education - English — The health education condition is a weekly 2-hour, 6 session course aimed at knowledge acquisition in subjects related to health care in general (in English)
  Arms: Health Education English
Behavioral: Health Education - Spanish — The health education condition is a weekly 2-hour, 6 session course aimed at knowledge acquisition in subjects related to health care in general (in Spanish)
  Arms: Health Education Spanish

SUMMARY:
This study explores the differential efficacy of Spanish or English versions of a mindfulness intervention on Depression levels, using a pre test post test design and an active control condition (health education).

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) with an experimental condition (MAPs Mindfulness intervention) and an active control group (Health Education), using a pretest and immediate posttest research design. Both conditions are comprised of a 6-week group intervention, which will be administered at the UCLA Westwood Medical Campus. The sample (N=80) will be drawn from a population of adults (18-65 years old), residing within a 10mile radius of the UCLA Westwood Medical Campus. To determine initial eligibility, potential participants will self-select based on perceived high levels of stress. Participants will respond self-report questionnaires to assess for psychological symptoms and will be drawn blood samples (180ml total) to assess levels of pro inflammatory cytokines before and after the interventions. Participants will attend a total of 8 visits.

ELIGIBILITY:
Inclusion Criteria:

* In order to determine eligibility, interested participants will be phone screened. To qualify for the study, participants have to be fluent in either Spanish or English, validated by self-report at phone screening. Additionally, during the phone screening participants had to complete a 4-item version of the Perceived Stress Scale (Cohen & Williamson, 1988) and score above the 50th percentile (a score of 9 or higher) in order to be eligible

Exclusion Criteria:

* People not meeting any of the above criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 6 weeks
  The Beck Depression Inventory (BDI) is a 21-item self-reporting questionnaire for evaluating the severity of depression in normal and psychiatric populations

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire | 6 weeks
  This instrument is based on a factor analytic study of five independently developed mindfulness questionnaires. The analysis yielded five factors that appear to represent elements of mindfulness as it is currently conceptualized. The five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.
Perceived Stress Scale | 6 weeks
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Higher scores represent overall higher levels of perceived stress. Scores range from 0 to 40 points.
Self Compassion Scale | 6 weeks
  The Self-Compassion Scale is a psychometrically sound and theoretically valid measure of self-compassion. Scores range from 26 to 130, with higher scores representing higher levels of self-compassion. All subscales (Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness and Over-identified) are combined to compute a total score.
Positive and Negative Affect Schedule | 6 weeks
  he Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Scores range from 10 to 50 points, with higher scores representing higher levels of positive or negative affect.
IL6 | 6 weeks
  Plasma concentrations of Interleukin-6
TNFa | 6 weeks
  Plasma concentrations of tumor necrosis factor alpha

REFERENCES:
- [Derived] Lopez-Maya E, Olmstead R, Irwin MR. Mindfulness meditation and improvement in depressive symptoms among Spanish- and English speaking adults: A randomized, controlled, comparative efficacy trial. PLoS One. 2019 Jul 5;14(7):e0219425. doi: 10.1371/journal.pone.0219425. eCollection 2019. PMID 31276540